CLINICAL TRIAL: NCT01387464
Title: A Double-Masked Clinical Study To Determine The Aqueous Humor Concentration Of Bromfenac Sodium In Subjects Administered Multiple Topical Ocular Doses Of ISV-303 Or Bromday™ Once Daily (QD) Prior To Cataract Surgery
Brief Title: Aqueous Humor Concentration of InSite Vision (ISV) 303 (Bromfenac in DuraSite) to Bromday Once Daily (QD) Prior to Cataract Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-11-303-002
Record Dates: First submitted 2011-06-29; First posted 2011-07-04 (Estimated); Results first posted 2016-06-02 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cataract
Keywords: bromfenac concentrations; ISV-303; Bromday
MeSH Terms: conditions — Cataract | interventions — bromfenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISV-303 (Experimental)
  Interventions: Drug: ISV-303
- Bromday™ (Active Comparator)
  Interventions: Drug: Bromday™

INTERVENTIONS:
Drug: ISV-303 — 0.075% bromfenac in DuraSite dosed QD
  Arms: ISV-303
Drug: Bromday™ — 0.09% bromfenac dosed QD
  Arms: Bromday™

SUMMARY:
The purpose of this study is to evaluate the aqueous humor concentration of bromfenac sodium in subjects administered multiple topical ocular doses of ISV-303 or Bromday™ QD prior to routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 or older scheduled for unilateral cataract surgery (phacoemulsification or extracapsular extraction) with posterior chamber intraocular lens implantation
* If a female is of childbearing potential, the subject must agree to and submit a urine sample for pregnancy testing at Visit 1 prior to enrollment and at the end of the study, and the subject must use effective contraception for the duration of the study. Post menopausal is defined as having no menses for at least 12 consecutive months.
* Signature of the subject on the Informed Consent Form
* Willing and able to follow all instructions and attend all study visits
* Able to self-administer study drug (or have a caregiver available to instill all doses of study drug)

Exclusion Criteria:

* Use of any drug containing bromfenac within 2 weeks prior to surgery
* Contact lens wear during the dosing period
* Known hypersensitivity or poor tolerance to bromfenac sodium or any component of the investigational medicinal product (IMP) or any of the procedural medications
* Any serious complications with or macroscopic damage to the corneal epithelium
* Currently pregnant, nursing, or planning a pregnancy; or be a woman that has a positive urine pregnancy test
* Currently suffer from alcohol and/or drug abuse
* Prior participation in this study protocol
* Prior (within 30 days of beginning study treatment) or anticipated concurrent use of an investigational drug or device
* A condition or a situation, which in the investigator's opinion may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- ISV-303: 0.075% bromfenac in DuraSite vehicle dosed QD
- Bromday: 0.09% bromfenac dosed QD
Period: Overall Study
Arm/Group | ISV-303 | Bromday
Started | 30 | 30
Safety Population | 30 | 29
Per-Protocol Population | 29 (Safety subjects who completed surgery) | 29
Completed | 29 | 29
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-303 | Bromday | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (10.14) | 68.2 (9.5) | 69.4 (9.8)
Age, Customized [Number; unit: participants]
  18-30 years | 0 | 0 | 0
  31-50 years | 1 | 0 | 1
  51-70 years | 10 | 18 | 28
  >70 years | 19 | 12 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 19 | 31
  Male | 18 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Aqueous Humor Bromfenac Concentration
Time Frame: Approximately 3 hours post last dose
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ISV-303 | Bromday
Number analyzed (Participants) | 29 | 29
ng/mL | 49.3 (41.87) | 23.7 (16.31)

ADVERSE EVENTS:
Time Frame: 4 days
Arm/Group | ISV-303 | Bromday
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other